CLINICAL TRIAL: NCT06453434
Title: The Impact of Continuous Glucose Monitoring Based Self-management on Patient-Reported Outcomes and Glycaemia in Type 1 Diabetes
Brief Title: Diabetes Self-management With Continuous Glucose Monitoring
Acronym: DIASELF
Status: Not yet recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1306-6133
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes
Keywords: Continuous Glucose Monitoring; Self-management; Diabetes Technology; Type 1 Diabetes; Diabetes Distress; Patient-reported Outcomes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this observational study is to investigate the interaction between people with type 1 diabetes and continuous glucose monitoring (CGM) and the impact of this interaction on quality of life, particularly the level of diabetes distress, and glycaemic metrics.

Participants will:

* Visit the clinic twice with a 14-day interval
* Fill out a survey before the first and at the last visit
* Use CGM as usual and use smart insulin pens and an activity tracker
* Register food intake
* Answer two-three questions twice a day in REDCap

DETAILED DESCRIPTION:
A two-centre observational study conducted in Denmark, including adults with type 1 diabetes (n=500) on multiple daily injections already using FreeStyle Libre 2.

Upon recruitment, participants will complete a survey of 11 validated questionnaires, including T1-DDS-28. For 14 days, participants will continue regular CGM use, smart insulin pens will record real-time insulin dosage, and an activity sensor will monitor physical activity and sleep. Participants will register food intake in the LibreLink app and respond to queries on quality of life twice daily through REDCap. At the end of the study, participants will complete the T1-DDS-28 and Health Literacy Questionnaire.

Our primary objectives is to investigate the association between diabetes distress (assessed by Type 1 Diabetes Distress Scale (T1-DDS-28)) and:

1. frequency of reading CGM data,
2. frequency of low glucose alarms,
3. frequency of high glucose alarms,
4. frequency of daily between-meal insulin corrections,
5. frequency of hypoglycaemic events preceded by correction of hyperglycaemia with insulin,
6. frequency of hyperglycaemic events preceded by correction of hypoglycaemia with carbohydrates, and
7. sociodemographic and psychosocial characteristics of CGM users.

Our secondary objective is to investigate the association between glycaemic metrics and the variables described above. Glycaemic metrics will be reported as CGM-metrics, including time in range defined as the percentage of time the sensor glucose is 3.9-10.0 mmol/L (70-180 mg/dL), per international consensus (ATTD, 2022)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years.
2. Diagnosed with T1D over one year ago.
3. Actively using FreeStyle Libre 2 (>80% sensor activity).
4. Used FreeStyle Libre 2 for over three months.
5. Uses multiple daily insulin injections.
6. Capable of providing written informed consent.
7. Willing and able to complete study procedures, including using smart caps or pens and completing questionnaires at the investigator's discretion.

Exclusion Criteria:

1. History of allergic reactions to materials or adhesives used in CGM devices.
2. Presence of severe cognitive or psychiatric conditions that could hinder the effective use of CGM or smart caps or pens - at the investigator's discretion.
3. Current use of steroids unless part of a chronic therapy plan.
4. Daily consumption of vitamin C ≥ 500 mg.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 1 diabetes (n=500) on multiple daily insulin injections already using FreeStyle Libre 2.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | At baseline and after 14 days.
  Type 1 Diabetes Distress Scale (T1-DDS-28)) Score. Likert scale. Score from 1 to 5. Higher scores indicate higher grade of diabetes distress.

SECONDARY OUTCOMES:
Time in range (TIR) | 14 days
  Time in range defined as the percentage of time the sensor glucose is 3.9-10.0 mmol/L (70-180 mg/dL)
Time in tight range (TIR) | 14 days
  The percentage of time the sensor glucose is 3.9-7.8 mmol/L (70-140 mg/dL)
Time below range level 1 (TBR1) | 14 days
  The percentage of time the sensor glucose is 3.0-3.9 mmol/L (54-70 mg/dL)
Time below range level 2 (TBR2) | 14 days
  The percentage of time the sensor glucose is <3.0 mmol/L (<54 mg/dL)
TBR1 night | 14 days
  TBR 3.0-3.9 from 0000h to 0559h, level 1 night
TBR1 day | 14 days
  TBR 3.0-3.9 from 0600h to 2359h, level 1 day
TBR2 night | 14 days
  TBR <3.0 from 0000h to 0559h, level 2 night
TBR2 day | 14 days
  TBR <3.0 from 0600h to 2359h, level 2 day
Time above range level 1 (TAR1) | 14 days
  The percentage of time the sensor glucose is 10.1-13.9 mmol/L (181-250 mg/dL)
Time above range level 2 (TAR2) | 14 days
  The percentage of time the sensor glucose is 13.9 mmol/L (>250 mg/dL)
TAR1 night | 14 days
  TAR1 10.1-13.9 from 0000h to 0559h, level 1 night
TAR1 day | 14 days
  TAR1 10.1-13.9 from 0600h to 2359h, level 1 day
TAR2 night | 14 days
  TAR2 >13.9 from 0000h to 0559h, level 1 night
TAR2 day | 14 days
  TAR2 >13.9 from 0600h to 2359h, level 1 day
Coefficient of variation (CV) | 14 days
  Measure of glucose variability. Calculated as 100 x (SD divided by mean glucose)
Mean sensor glucose | 14 days
  Mean sensor glucose (mmol/L and mg/dL)
Standard deviation of mean glucose (SD) | 14 days
  Standard deviation of mean glucose (SD) (mmol/L and mg/dL)

OTHER OUTCOMES:
Frequency of daily CGM readings | 14 days
  How many times the participants open the LibreView app to assess their CGM data during the day
Diurnal variation of daily CGM readings | 14 days
  Numbers in the morning (06.00-11.59), afternoon (12.00-17.59), in the evening (18.00-23.59) and in the night (00.00-05.59)
Active sensor | 14 days
  Percentage of sensor data obtained
Frequency of daily between-meal insulin corrections | 14 days
  How many times the participants take between-meal insulin corrections daily
Frequency of hypoglycaemic events preceded by correction of hyperglycaemia with insulin, | 14 days
  For each hypoglycaemic event (defined as a glucose level ≥ 10 mmol/L (180 mg/dL)) a cause of the event will be interpreted based on 4-hours data and classified as either preceded by 1) premeal-insulin, 2) insulin correction of hyperglycemia or 3) physical activity
Frequency of hyperglycaemic events preceded by correction of hypoglycaemia with carbohydrates | 14 days
  For each hyperglycaemic event (defined as glucose level ≥ 10 mmol/L (180 mg/dL) ≥ 15 consecutive minutes) a cause of the event will be interpreted based on 4-hours data and classified as either preceded by 1) carbohydrate intake without premeal insulin, 2) carbohydrate intake with premeal insulin, or 3) correction of hypoglycaemia with carbohydrate
High glucose alarm threshold | At baseline
  Mean/median alarm threshold level at baseline
Low glucose alarm threshold | At baseline
  Mean/median alarm threshold level at baseline
Frequency of high glucose alarms | 14 days
  Number of high glucose alarms during the study
Frequency of low glucose alarms | 14 days
  Number of low glucose alarms during the study
Low alarms enabled | 14 days
  Percentage of time low alarms are activated
High alarms enabled | 14 days
  Percentage of time high alarms are activated
Diurnal variation of high alarms | 14 days
  Numbers in the morning (06.00-11.59), afternoon (12.00-17.59), evening (18.00-23.59) and night (00.00-05.59)
Diurnal variation of low alarms | 14 days
  Numbers in the morning (06.00-11.59), afternoon (12.00-17.59), evening (18.00-23.59) and night (00.00-05.59)
Smart pen engagement | 14 days
  Number of days with data uploads during the study period
Total daily dose (TDD) of insulin | 14 days
  Mean of the study period. Recorded by smartpens.
Total daily dose (TDD) of basal insulin | 14 days
  Mean of the study period. Recorded by smartpens.
Total daily dose (TDD) of insulin delivered as premeal boluses | 14 days
  Mean of the study period. Recorded by smartpens.
Total daily dose (TDD) of insulin delivered as correctional boluses | 14 days
  Mean of the study period. Recorded by smartpens.
Percentage of TDD of insulin delivered as correctional boluses out of TDD of insulin | 14 days
  Percentage
Missing basal insulin dose | 14 days
  ≥ 40 hours between basal insulin injections
Missing meal boluses | 14 days
  No bolus injection within 15 minutes before and 60 minutes after the start of a meal. Meals identified using a food diary/CGM signal by using the GRID algorithm.
Diurnal variation of correctional boluses | 14 days
  Numbers in the morning (06.00-11.59), afternoon (12.00-17.59), in the evening (18.00-23.59) and in the night (00.00-05.59), respectively
Step count per day | 14 days
  From activity sensor
Moderate and vigorous physical activity (MVPA) | 14 days
  From activity sensor. Time spent on moderate and vigorous physical activity (MVPA)
Low-intensity physical activity (LPA) | 14 days
  From activity sensor. Time spent on low-intensity physical activity (LPA) time
Total physical activity (TPA) level | 14 days
  From activity sensor. TPA measured in counts per minute
Sleep | 14 days
  From activity sensor. Sleep hours per night
Food intake | 14 days
  Database which contains food intake data (amount of food in carbohydrates) retrieved from the diary app (LibreLink).
Food intake | 14 days
  Database which contains food intake data (timing of food intake) retrieved from the diary app (LibreLink).
Clarke score | At baseline
  Patient-reported outcome regarding awareness of hypoglycemia.
Gold score | At baseline
  Patient-reported outcome regarding awareness of hypoglycemia.
Hilleroed method | At baseline
  Patient-reported outcome regarding awareness of hypoglycemia.
Glucose Monitoring Satisfaction Survey (GMSS) | At baseline
  Patient-reported outcome regarding CGM satisfaction
Perceived Competence in Diabetes (PCD) | At baseline
  Patient-reported outcome regarding diabetes self-management
Diabetes Treatment Satisfaction Questionnaire status (DTSQs) | At baseline
  Patient-reported outcome regarding diabetes treatment satisfaction
Hypoglycaemia Fear Survey-II Short Form (HFS-SF) | At baseline
  Patient-reported outcome regarding fear of hypoglycemia
The Danish Health Literacy Questionnaire (HLQ) | At baseline
  Patient-reported outcome regarding health literacy
Based on Saltin-Grimby Physical Activity Level Scale (SGPALS) | At baseline
  Patient-reported outcome regarding physical activity
Well-Being Index (WHO-5) | At baseline
  Patient-reported outcome regarding psychological well-being
Pittsburgh Sleep Quality Index (PSQI) | At baseline
  Patient-reported outcome regarding sleep quality
Type D scale (DS-14) | At baseline
  Patient-reported outcome regarding type D personality trait
VAS-A | Each morning and each evening during the study period
  Patient-reported outcome regarding anxiety
EQ-VAS | Each morning during the study period
  Patient-reported outcome regarding overall health

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Pedersen-Bjergaard, Professor, Principal Investigator — Copenhagen University Hospital, North Zealand - Hollered
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Herlev, Capital Region
  - Copenhagen University Hospital, North Zealand - Hilleroed, Hillerød, Capital Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nitschke MJ, Demir C, Brosen JMB, Tapager IW, Norgaard K, Kristensen PL, Pedersen-Bjergaard U. Diabetes self-management observational study investigating how CGM use impacts diabetes distress, glycaemia and functions as a technological substitute for hypoglycaemia awareness: a study protocol. BMJ Open. 2025 Sep 2;15(9):e103469. doi: 10.1136/bmjopen-2025-103469. PMID 40897486